CLINICAL TRIAL: NCT03797859
Title: Apneic Oxygenation With Transnasal Humidified Rapid Insufflation Ventilatory Exchange (THRIVE) With Standardized Airway Management During General Anesthesia - an Observational Study of Blood Gas Dynamics of PaCO2, pH and PaO2.
Brief Title: THRIVE Apneic Ventilation With Standardized Airway Management During General Anesthesia.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Seltz Kristensen, SENIOR CONSULTANT, Rigshospitalet, Denmark
Other Study IDs: H-18017844
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Apnea; Ventilation Therapy; Complications; Respiratory Acidosis
MeSH Terms: conditions — Apnea; Acidosis, Respiratory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Apneic ventilation — Ventilation by THRIVE

SUMMARY:
Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) denotes the use of high-flow humidified nasal oxygen system (for example Optiflow®) as an alternative ventilation modality for an anesthetized patient without spontaneous respiration. This method requires only basic airway management manoeuvres to keep the airway open and provides both stable longterm oxygenation as well as apneic ventialtion.

We plan to evaluate this methods physiological performance under standardized conditions of airway management by frequent, repeated arterial blood gas analyses.

DETAILED DESCRIPTION:
THRIVE is previously shown feasible as sole mode of ventilation in selected patients during general anaesthesia for minor laryngeal surgery for a limited time up to 30 minutes, where direct laryngoscopy was required and applied throughout the procedure. A stable oxygenation and a degree of ventilation was observed. However, a slowly developed respiratory acidosis was also observed over time.

Existing physiologic studies on high flow humidified nasal oxygen suggest that closed mouth breathing enhance the effects of the high flows of oxygen levels applied by increasing the airway pressures and thereby enhance gas exchange in the lungs. Currently, it is unclear whether the efficiency of THRIVE depends on the particular circumstances of airway management. Physiologic characterization of THRIVE performance under standardized conditions of airway management and under close monitoring by systematic analysis of blood gas dynamics over time during general anesthesia is needed.

We plan to study the blood gas dynamics during THRIVE apnea ventilation during general anesthesia, where the airway is managed only by jaw-thrust for up to 60 minutes. The patients will be closely monitored by repetitive arterial blood gasses to evaluate blood gas dynamics and development of respiratory acidosis. Desaturation or respiratory acidosis with pH under 7.15 and/or PaCO2-rise > 12 kPa will lead to cessation of THRIVE.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age over 18 years)
2. Elective surgery where intubation is not mandatory
3. The patient can understand the information about the study and give their informed written consent of participation

Exclusion Criteria:

1. ASA (American Society of Anaesthesiologists class) > 3
2. NYHA (New York Heart Association class) > 2
3. BMI > 30 kg/m2
4. Symptomatic respiratory disease
5. Symptomatic cardiac disease
6. Evidence of arteriosclerotic disease
7. Neuromuscular disease
8. Pregnancy
9. Presumed or predicted difficult airway (SARI - Simplified Airway Risk Index score > 4)
10. Known or suspected nasal congestion/stenosis or catharalia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting for non-laryngeal surgery in general anesthesia, where intubation is not mandatory.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory acidosis | Max. 60 minutes
  Development of respiratory acidosis (pH < 7.15 or paCO2 > 12) over time on study

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Kristensen, MD, Principal Investigator — Senior consultant, Rigshospitalet
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen, Hoevdstaden
  - Rigshospitalet, section for anaesthesia for ENT and Maxillofacial surgery, section 3071, Copenhagen

IPD SHARING:
Plan to Share IPD: No